CLINICAL TRIAL: NCT05506982
Title: The Safety, Feasibility, and Acceptability of Psilocybin Combined With Multidisciplinary Palliative Care in Demoralized Cancer Survivors With Chronic Pain (P-PC)
Brief Title: Psilocybin Combined With Multidisciplinary Palliative Care in Demoralized Cancer Survivors With Chronic Pain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ali Zarrabi, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00001905; NCI-2020-13913 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00001905 (Other: Emory University Hospital/Winship Cancer Institute); EU5206-20 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-08-06; First posted 2022-08-18 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Psilocybin; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Supportive care (psilocybin, observation) (Experimental): Patients receive psilocybin PO and undergo observation for up to 24 hours on day 14.
  Interventions: Drug: Psilocybin; Behavioral: Psychotherapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Psilocybin — Given PO
  Other Names: CY-39; Indocybin
Behavioral: Psychotherapy — supportive care
  Other Names: talk therapy
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase I trial evaluates the side effects of psilocybin and how well it works under supportive care conditions in cancer survivors living with demoralization and chronic pain. Cancer patients often experience demoralization, which is characterized by feelings of hopelessness, loss of meaning, and existential distress. Psilocybin psychotherapy, together with multidisciplinary palliative and supportive care, may help treat the anxiety, depression, and chronic pain felt by cancer survivors - defined here as cancer patients from time of diagnosis through the end-of-life.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety, feasibility, and acceptability of a single administration of 25 mg psilocybin (psilocybin) provided under supportive conditions with multidisciplinary palliative care support (P-PC) in adult cancer survivors living with concurrent demoralization and chronic pain.

EXPLORATORY OBJECTIVE:

I. To evaluate for changes in demoralization, anxiety, depression, quality of life, pain, other symptoms, mysticism, awe, post-traumatic growth, social isolation, and psychosocial functioning from baseline to end-of-treatment to 3.5-month follow up.

OUTLINE:

Patients receive psilocybin orally (PO) and undergo observation for up to 8 hours on day 14.

After completion of study intervention, patients are followed up on days 15, 21, 42, 56, and 98.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF)
* Diagnosis of solid or liquid cancer made >= 1 year at any stage in cancer survivorship (specifically, active cancer treatment or no cancer-directed therapy either in clinical remission or with advanced disease)
* Prognosis of greater than six months as determined by their primary oncologist
* Moderate-to-severe demoralization (score of >= 10 on the Demoralization Scale-II [DS-II])
* Chronic pain (pain lasting > 3 months) per patient report and score of >= 5 for average pain level on Brief Pain Inventory
* Age >= 26 years old and ≤85 years old
* Availability of a friend or family member into whose care the participant can be released following the drug administration session

Exclusion Criteria:

* Pregnancy or breastfeeding
* Women of childbearing potential (i.e., not permanently sterilized, not postmenopausal) who decline to use a highly effective dual contraceptive method for the duration of the study. Dual contraceptive method use is defined by a use a barrier contraceptive in addition to another method to prevent pregnancy, including sterilization, hormonal methods, intrauterine devices, and hormonal pills.
* Age < 26 years old and > 85 years old
* Poor functional status (Eastern Cooperative Oncology Group [ECOG] score of >= 2)
* Major cognitive impairment as determined by principal investigator
* Non-fluency in the English language
* Personal history of a psychotic disorder or Bipolar disorder type I/II
* Active suicidal ideation with intent in the last 3 months (Columbia Suicide Severity Rating Scale suicidal ideation score > 3) or any suicide attempt in the past year
* Current substance use disorder (i.e., present in last six months), of greater than mild severity as defined by Diagnostic and Statistical Manual of Mental Disorders (DSM-V)
* History of a seizure disorder in adulthood
* Active central nervous system (CNS) metastases or symptomatic CNS infection
* Uncontrolled hypertension (mean blood pressure (mmHg) exceeding 139 systolic and 89 diastolic) and heart rate exceeding 90 beats per minute
* Clinically significant cardiovascular disease (coronary artery disease, congestive heart failure, arrhythmia, or QTc>450ms)
* Supplemental oxygen requirement
* Body mass index =< 18
* Renal insufficiency as evidenced by creatinine clearance (CrCl) < 30 mL/min
* Concomitant use of drugs known to interact with psilocybin (probenecid, diclofenac)
* Consistent use of serotonergic drugs including selective serotonin reuptake inhibitors (SSRIs), serotoninnorepinephrine reuptake inhibitors (SNRIs), or efavirenz, as well as monoamine oxidase inhibitors (MAOIs). Subjects using any other antidepressant, stimulant, or antipsychotic medications on Day 0 (baseline visit) may be allowed to enroll in the study if they elect to taper off the medications under medical supervision by the PI and the study psycho-oncologist (PO) by the day prior to the baseline visit
* Considered by the principal investigator to be inappropriate for the study due to safety concerns or to be unlikely to complete the protocol

Min Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2024-04-25 (Actual); Study Completion 2025-01-24 (Actual)

PRIMARY OUTCOMES:
Incidence Of Treatment-Related Medical Grade 3 Or Higher Or Psychiatric Grade 4 Or Higher | Up to 42 days
  Adverse events are graded according to Common Terminology Criteria for Adverse Events. Descriptive statistics will summarize the incidence and duration of adverse events, with the primary outcome of interest being the incidence of medical Grade 3 or higher or psychiatric Grade 4 or higher Common Terminology Criteria for Adverse Events considered by the PI to be treatment-related occurring by day 42. These events will be evaluated by adverse events, vital signs, ECG, and laboratory findings. A successful outcome is no medical or psychiatric Grade 4 adverse events or higher.
Evaluation of Feasibility Outcome To Assess Patient Retention in The Study | Up to 42 days
  Feasibility will be assessed by patient retention in the study, number of missed events, a survey assessing acceptability of the protocol at study endpoint, and fidelity to the intervention elements. A successful outcome is retention of 80% of subjects enrolled in the study, 80% of events attended by subjects, and 60% of subjects find intervention satisfactory.

OTHER OUTCOMES:
Evaluate for Changes in Demoralization at Forty-Two Days | At 42 days
  Evaluate demoralization using the Demoralization Scale from baseline to end-of-treatment to 3.5-month follow up. Moderate-to-severe demoralization (score of ≥ 10 on the Demoralization Scale-II).
Evaluate for Changes in Demoralization at Ninety-Eight Days | At 98 days
  Evaluate demoralization using the Demoralization Scale from baseline to end-of-treatment to 3.5-month follow up. Moderate-to-severe demoralization (score of ≥ 10 on the Demoralization Scale-II).
Impact of Pain Intensity and Interference with Daily Functioning at Forty-Two Days | At 42 days
  The impact of pain intensity and interference with daily functioning will be assessed using Brief Pain Inventory. Chronic pain (pain lasting > 3 months per patient report) and score of ≥ 5 for average pain level on Brief Pain Inventor.
Impact of Pain Intensity and Interference with Daily Functioning at Ninety-Eight Days | At 98 days
  The impact of pain intensity and interference with daily functioning will be assessed using Brief Pain Inventory. Chronic pain (pain lasting > 3 months per patient report) and score of ≥ 5 for average pain level on Brief Pain Inventor.
Global Symptom Burden at Forty-Two Days | At 42 days
  Global symptom burden will be evaluated using the Edmonton Symptom Assessment Scale.The scale ranges from 0 representing no symptom to 10 representing maximum symptom.
Global Symptom Burden at Ninety-Eight Days | At 98 days
  Global symptom burden will be evaluated using the Edmonton Symptom Assessment Scale.The scale ranges from 0 representing no symptom to 10 representing maximum symptom.
Anxiety and Depression at Forty-Two Days | At 42 days
  Anxiety and Depression is evaluated using the Hospital Anxiety and Depression Scale.
  The Hospital Anxiety and Depression Scale is a 14-item self-report scale and reliable instrument for detecting states of depression and anxiety in outpatient settings, where 0-7 = Normal, 8-10 = Borderline abnormal (borderline case) and 11-21 = Abnormal (case).
Anxiety and Depression at Ninety-Eight Days | At 98 days
  Anxiety and Depression is evaluated using the Hospital Anxiety and Depression Scale.
  The Hospital Anxiety and Depression Scale is a 14-item self-report scale and reliable instrument for detecting states of depression and anxiety in outpatient settings, where 0-7 = Normal, 8-10 = Borderline abnormal (borderline case) and 11-21 = Abnormal (case).
Quality of Life Assessment at Forty-Two Days | At 42 days
  Evaluated quality of life changes from baseline to end-of-treatment to 3.5-month follow up using the Harvard Flourishing Measure. Life Satisfaction (Items 1-2) ranges from 0 = Not Satisfied at All, 10 = Completely Satisfied, Mental and Physical Health (3-4) ranges from 0 = Poor, 10 = Excellent, Meaning and Purpose (5-6) ranges from 0 = Not at All Worthwhile, 10 = Completely Worthwhile and 0 = Strongly Disagree, 10 = Strongly Agree, Character and Virtue (7-8) ranges from 0 = Not True of Me, 10 = Completely True of Me, and Close Social Relationships (9-10) ranges from 0 = Strongly Disagree, 10 = Strongly Agree. A sixth domain, Financial and Material Stability (11-12) may be necessary to sustain the other domains over time ranges from 0 = Worry All of the Time, 10 = Do Not Ever Worry.
  .
Quality of Life Assessment at Ninety-Eight Days | At 98 days
  Evaluated quality of life changes from baseline to end-of-treatment to 3.5-month follow up using the Harvard Flourishing Measure. Life Satisfaction (Items 1-2) ranges from 0 = Not Satisfied at All, 10 = Completely Satisfied, Mental and Physical Health (3-4) ranges from 0 = Poor, 10 = Excellent, Meaning and Purpose (5-6) ranges from 0 = Not at All Worthwhile, 10 = Completely Worthwhile and 0 = Strongly Disagree, 10 = Strongly Agree, Character and Virtue (7-8) ranges from 0 = Not True of Me, 10 = Completely True of Me, and Close Social Relationships (9-10) ranges from 0 = Strongly Disagree, 10 = Strongly Agree. A sixth domain, Financial and Material Stability (11-12) may be necessary to sustain the other domains over time ranges from 0 = Worry All of the Time, 10 = Do Not Ever Worry.
Caregiver strain at Forty-Two Days | At 42 days
  The Measured by the Modified Caregiver Strain Index is a 13-item tool measuring strain related to care provision with at least one item for each of the following major domains: financial, physical, psychological, social, and personal. The instrument is used to assess individuals of any age who assume the role of care giving.The index ranges from: Yes, On a Regular Basis=2, Yes, Sometimes =1, and No=0.
Caregiver strain at Ninety-Eight Days | At 98 days
  The Measured by the Modified Caregiver Strain Index is a 13-item tool measuring strain related to care provision with at least one item for each of the following major domains: financial, physical, psychological, social, and personal. The instrument is used to assess individuals of any age who assume the role of care giving.The index ranges from: Yes, On a Regular Basis=2, Yes, Sometimes =1, and No=0.
Impact of pain intensity and interference with catastrophizing through rumination, helplessness, and pessimism at Forty-Two Days | At 42 days
  Evaluated using the Pain Catastrophizing Scale. Where 0=Not at all, 1=To a slight degree, 2=To a moderate degree, 3=To a great degree, 4= All the time.
Impact of pain intensity and interference with catastrophizing through rumination, helplessness, and pessimism at Ninety-Eight Days | At 98 days
  Evaluated using the Pain Catastrophizing Scale. Where 0=Not at all, 1=To a slight degree, 2=To a moderate degree, 3=To a great degree, 4= All the time.
Religious and spiritual assessment at Forty-Two Days | At 42 days
  Evaluated using Santa Clara Strength of Religious Faith Questionnaire. 1 = strongly disagree, 2 = disagree, 3 = agree and 4 = strongly agree.
Religious and spiritual assessment at Ninety-Eight Days | At 98 days
  Evaluated using Santa Clara Strength of Religious Faith Questionnaire. 1 = strongly disagree, 2 = disagree, 3 = agree and 4 = strongly agree.
Social connectedness at Forty-Two Days | At 42 days
  Evaluated using the Social Connectedness Scale-Revised. The Social Connectedness Scale-Revised is a validated 8-item self-report measure assessing the degree to which subjects feel socially connected as a psychological sense of belonging. Where 1= Strongly Disagree, 2= Disagree, 3=Mildly Disagree, 4= Mildly Agree, 5= Agree, 6= Strongly Agree
Social connectedness at Ninety-Eight Days | At 98 days
  Evaluated using the Social Connectedness Scale-Revised. The Social Connectedness Scale-Revised is a validated 8-item self-report measure assessing the degree to which subjects feel socially connected as a psychological sense of belonging. Where 1= Strongly Disagree, 2= Disagree, 3=Mildly Disagree, 4= Mildly Agree, 5= Agree, 6= Strongly Agree
Self-reported opioid use in the form of oral morphine equivalents over past week at Forty-Two Days | At 42 days
  Opioid use in the form of oral morphine equivalents.
Self-reported opioid use in the form of oral morphine equivalents over past week at Ninety-Eight Days | At 98 days
  Opioid use in the form of oral morphine equivalents.
Self-reported polypharmacy over past week at Forty-Two Days | At 42 days
  The number of total medications used to manage physical and emotional symptoms
Self-reported polypharmacy over past week | At 98 days
  The number of total medications used to manage physical and emotional symptoms
Global psychosocial functioning (participant and caregiver) at Forty-Two Days | At 42 days
  Evaluated using using the Work and Social Adjustment Scale. It is a 5-item measure of general social impairment, and specifically their ability to function in terms of work, tasks at home, social leisure, private leisure, and personal or family relationships. Score: 0-9= low impairment, 10-19= moderate impairment, 20-40 severe impairment.
Global psychosocial functioning (participant and caregiver) at Ninety-Eight Days | At 98 days
  Evaluated using using the Work and Social Adjustment Scale. It is a 5-item measure of general social impairment, and specifically their ability to function in terms of work, tasks at home, social leisure, private leisure, and personal or family relationships. Score: 0-9= low impairment, 10-19= moderate impairment, 20-40 severe impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Ali J. Zarrabi, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (2):
- United States (2):
  - Emory University/Winship Cancer Institute, Atlanta, Georgia
  - Brain Health Center at Executive Park, Atlanta, Georgia